CLINICAL TRIAL: NCT02298400
Title: A Single-Center, Cross-over, Pilot Study Evaluating Acuvue® Oasys® Lenses (Senofilcon A), 30-Day Bausch + Lomb PureVision (Balafilcon A), and Clariti® 1-Day (Somofilcon A) Lenses, for Their Impact on Ocular Discomfort Induced by Exposure to the Turbo Controlled Adverse Environment™
Brief Title: A Clinical Study Comparing the Comfort of Three Commercially Available Contact Lenses
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated by Sponsor
Sponsor: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 14-270-0001
Record Dates: First submitted 2014-11-17; First posted 2014-11-24 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Contact Lens Complication

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acuvue®Oasys® Lenses(senofilcon A) (Active Comparator): Acuvue® Oasys® Lenses (senofilcon A) contact lenses
  Interventions: Device: Acuvue® Oasys® Lenses (senofilcon A); Device: 30-Day Bausch + Lomb PureVision (balafilcon A); Device: Clariti® 1-Day (Somofilcon A)
- Bausch + Lomb PureVision (balafilcon A) (Active Comparator): 30-Day Bausch + Lomb PureVision (balafilcon A) contact lenses
  Interventions: Device: Acuvue® Oasys® Lenses (senofilcon A); Device: 30-Day Bausch + Lomb PureVision (balafilcon A); Device: Clariti® 1-Day (Somofilcon A)
- Clariti® 1-Day (Somofilcon A) (Active Comparator): Clariti® 1-Day (Somofilcon A) contact lenses
  Interventions: Device: Acuvue® Oasys® Lenses (senofilcon A); Device: 30-Day Bausch + Lomb PureVision (balafilcon A); Device: Clariti® 1-Day (Somofilcon A)

INTERVENTIONS:
Device: Acuvue® Oasys® Lenses (senofilcon A) — Contact lenses placed in each eye during the day for about 8 hours
Device: 30-Day Bausch + Lomb PureVision (balafilcon A) — Contact lenses placed in each eye during the day for about 8 hours
Device: Clariti® 1-Day (Somofilcon A) — Contact lenses placed in each eye during the day for about 8 hours

SUMMARY:
The purpose of this study is to compare the comfort of three commercially available contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old
* Have provided written informed consent
* Have discomfort when wearing contact lenses

Exclusion Criteria:

* Have an active ocular infection or significant slit lamp findings
* Participated in any other studies in the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Contact lens wear comfort, as assessed by subject reported symptoms in diaries. | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States